CLINICAL TRIAL: NCT01245829
Title: Bacterial Contamination of Critical Care Observation Charts: a Randomized Trial Comparing Matt and Antimicrobial Cellomed Laminates.
Brief Title: A Randomized Trial Comparing Matt and Antimicrobial Cellomed Laminates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: County Durham and Darlington NHS Foundation Trust (Other Government)
Responsible Party: Dr Richard Hixson, County Durham and Darlington NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Cellomed001
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Cross Infection; Infection Control
Keywords: Cross Infection; Nosocomial Infection; Healthcare Acquired Infection; Hospital Paperwork; Observation Charts; Critical Care; Contamination
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matt (Placebo Comparator): A standard non antimicrobial laminated chart which will form the control group (group 1).
  Interventions: Other: Swabbing of observation chart
- Cellomed (Experimental): Observation charts coated in a laminate with antimicrobial properties (Cellomed) will form group 2.
  Interventions: Other: Swabbing of observation chart

INTERVENTIONS:
Other: Swabbing of observation chart — The observation charts to be studied will be stored on the DMH critical care unit and all existing non-laminated white charts removed for the duration of the study period. The observation charts will thereafter be used in the normal way as defined by nursing practice; blue charts from patient admission (irrespective of time) and white charts for each 24 hour period thereafter commencing at 8 am. On placement and after 24 hours of use, a standardised section of the patient observation area will be swabbed by the data collection researcher. The standardised area is defined as the section of the chart that is most comprehensively completed during the patient episode and is therefore most likely to become contaminated through contact. Use of white charts only is required in order to standardise the length of time each chart is in place between the two points of swabbing (white charts present at 8 am have been in use for exactly 24 hours).

SUMMARY:
Sepsis contributes to nearly 20% of all hospital deaths and is the leading cause of death on non-coronary intensive care units. Contamination of the patient environment is common with organisms such as MRSA, VRE and C.difficile remaining viable for days or weeks on a variety materials and surfaces. Up to 90% of patient notes and charts on critical care may be contaminated with potential pathogens including MRSA and it has been shown that healthcare workers may contaminate hospital paperwork with organisms originating from patients. Cellomed is a triclosan based laminate which has been shown to possess antimicrobial activity against MRSA, E.Coli, Enterococcus, Stenotrophomonas and Klebsiella. The study presented for consideration aims to compare levels of contamination between critical care observation charts coated with either a 'standard' matt or antimicrobial Cellomed laminate. It is proposed that paperwork laminated with Cellomed may exhibit reduced levels of contamination and decrease the potential for cross infection on critical care and potentially other areas of the hospital in which clinical paperwork is handled.

DETAILED DESCRIPTION:
Although hand hygiene remains an important intervention in reducing the incidence of nosocomial infection, poor compliance may limit its impact especially in critical care units when clinical demands on staff are high. Although focused programmes to improve compliance have been shown to produce good results this may not be sustained in the longer-term. Hand hygiene only reduces and does not completely eliminate hand contamination and therefore transmission of hand microbes to the near-patient environment including paperwork will inevitably occur. It is recommended that healthcare professionals undertake hand hygiene after interacting with the patient environment even if contact with the patient has not taken place. In practice this may not occur as the potential for the environment to act as a reservoir may not be realised by healthcare workers.

Doctors reviewing physiological trends on critical care observation charts often move between bed-spaces without touching patients or undertaking hand hygiene. Since doctors exhibit the lowest level of compliance with hand hygiene programmes, it is likely to be difficult to persuade them to undertake additional manoeuvres before and after handing paperwork as has been recommended. Effective cleaning and disinfection of the near-patient environment should occur concurrently to hand hygiene programmes in order to reduce transmission. Critical care observation charts in Darlington Memorial Hospital are paper-based, located in near-patient hand-touch zones and are therefore prone to contamination. It is proposed that treated paperwork may exhibit reduced levels of contamination; decreasing the potential for cross infection resulting from an area of the near-patient hand-touch environment that has received little attention in the past.

Recently published research (2009) has reported that up to 90% of critical care observation charts may be contaminated with potential or actual pathogens. It is on critical care where nosocomial infections potentially have the most devastating effect. Cellomed is a triclosan based laminate that has been available since 2008 through Celloglas, a UK company specialising in decorative and other print finishes. Celloglas claim the laminate possesses anti-microbial activity citing three reports from Ciba laboratories (Switzerland), Scientific Services (UK) and Manchester University (UK). All tests have shown activity against MRSA and E.Coli with the most recent test reporting additional activity against Enterococcus, Stenotrophomonas and Klebsiella when compared to control. To date there have been no studies of Cellomed carried out in the clinical environment. Cellomed can be applied to any hospital paperwork through a lamination process. It is proposed that 'treated' paperwork will exhibit reduced levels of contamination when used in the clinical environment compared with standard patient documentation.

This will be a prospective, randomised study comparing percentage increases in bacterial total viable count on critical care observation charts coated with one of two different materials; standard matt or Cellomed antibacterial laminate.

Two-hundred of our standard white critical care observation charts will be provided to Celloglas (Leeds, UK). 100 of these will be laminated with standard matt (group 1) and 100 with anti-microbial Cellomed (group 2). The two types of charts will be separately packaged by Celloglas, labelled and delivered to lead investigator at Darlington Memorial Hospital. The packages will be opened on a sterile work surface and the lead investigator will number the charts in a random order determined by an Excel spreadsheet. Randomisation will be restricted to ensure 100 charts remain in each group. The lead investigator will record which chart type is assigned to each number for analysis purposes. The charts will be used by the critical care nursing staff in the assigned order to ensure the random sequence is maintained.

The observation charts to be studied will be stored on the critical care unit and all existing non-laminated white charts removed. The observation charts will thereafter be used in the normal way as defined by nursing practice; blue charts for patient admissions and white charts for each 24 hour period thereafter commencing at 8 am. On placement and after 24 hours of use, a standardised section of the patient observation area will be swabbed by one of the data collection researchers. The standardised area is defined as the section of the chart that is most comprehensively completed during the patient episode and is therefore most likely to become contaminated through use. Both data collection researchers will be fully aware of the standardised area prior to commencement of the study.

White charts are used to standardise the length of time each chart is in place between pre- and post- clinical use swabs (white charts present at 8 am have been in use for exactly 24 hours). Blue charts are used between patient admission and 8 am which is a variable length of time and therefore not suitable for analysis.

All swabs will be taken by one of two data collection researchers using a standard technique agreed before data collection commences. One dry sterile cotton swab will thoroughly sample the specified area of white charts at 8 am. These charts will have been in use for 24 hours and therefore the swab casing will be marked with the chart identifying number, bed space number and the word 'post'. A new white patient observation chart will then be placed in the bed space by nursing staff and the same area swabbed using an identical method. The swab casing will be marked with the chart identifying number, the bed space number and the word 'pre'. Over a 24 hour period, each chart will therefore have two swabs taken; one pre- and one post- clinical use. The only exception to this will be on the first and the last day of the study when only pre- and post- swabs will be taken respectively.

Swabs will be immediately delivered to the laboratory and inoculated onto 'plates' to permit bacterial and fungal growth. Following 24 hours of incubation at 37 degrees Celsius in air, plates will be analysed for total viable count and specific bacteria identified using standard techniques within our accredited microbiology laboratory. Additional analysis for resistance of isolated Staphylococcus aureus and Enterococci will take place using British Society of Antimicrobial Chemotherapy (BSAC) standard techniques. All data relating to total viable counts and specific bacteria will be retained by the Data Collection Researchers until the study period has been concluded. No interim data will be generated.

The objectives are to compare the two groups total viable counts following 24 hours of clinical use and to compare the number of separately identified organisms. Unpublished laboratory tests show that total viable counts increases with manual handling of either laminate and it is therefore assumed that TVCs will increase from baseline for both types of observation chart following 24 hours of clinical use. Due to the claimed continuous expression of antimicrobial activity, there is the potential for baseline counts to be lower in the Cellomed group on receipt from the lamination factory. In addition, it cannot be assumed that the baseline contamination will be identical for charts between or within the two groups. It is therefore proposed to define the primary outcome measure as the percentage increase in total viable count from pre- 24 hour levels as measured before clinical use. The null hypothesis for the primary outcome measure is that there will be no difference in the percentage increase from baseline for total viable counts between the two groups following 24 hours of clinical use on the critical care unit. The alternative hypothesis is that Cellomed laminate results in a lower percentage increase in bacteria compared to standard matt laminate. The secondary outcome measure is to compare the number of different types of specific organisms identified during the laboratory analysis. The null hypothesis for the secondary outcome is that there will be no difference in the number of different types of specific organisms between the two groups following 24 hours of clinical use on the critical care unit. The alternative hypothesis is that Cellomed laminate results in fewer different types of specific organisms compared to standard matt laminate.

ELIGIBILITY:
Inclusion Criteria:

* All 200 of the specifically prepared, laminated white observation charts present on critical care will be included in the study.

Exclusion Criteria:

* White critical care charts in place at the time of a patient discharges will be excluded from analysis. This is due to the fact they would not have been in place for the full 24 hours and would not be available to have the 2nd swab sample taken. Blue observation charts are excluded since they are used for a variable period of time between patient admission and 8 am.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Percentage increase in bacteria total viable count | 24 hours
  Due to the claimed continuous expression of antimicrobial activity, there is the potential for baseline total viable counts to be lower in the Cellomed group on receipt from the lamination factory. In addition, it cannot be assumed that the baseline contamination will be identical for charts between or within the two groups. It is therefore proposed to define the primary outcome measure as the percentage increase in total viable count from pre- 24 hour levels as measured before clinical use on critical care.

SECONDARY OUTCOMES:
To compare the number of different types of specific organisms identified during the laboratory analysis. | 24 hours
  The secondary objective is to compare the number of different types of specific organisms identified in the two groups following 24 hours of clinical use.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Hixson, FRCA, Principal Investigator — County Durham and Darlington Acute Hospitals NHS Foundation Trust
Locations (1):
- Darlington Memorial Hospital, Darlington, County Durham, United Kingdom